CLINICAL TRIAL: NCT02844959
Title: Assessment of Course of Inflammatory Biomarkers Concentrations After Pulmonary Veins Isolation as a Prognostic Factor of Atrial Fibrillation Treatment Effectiveness (ACtIVE-AF Study)
Brief Title: Inflammatory Response as a Prognostic Factor of Recurrence of Atrial Fibrillation After Ablation
Acronym: ACtIVE-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marcin Grabowski, Clinical Professor, Marcin Grabowski, Medical University of Warsaw, Medical University of Warsaw
Other Study IDs: KB/143/2016
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Biomarkers; Inflammatory Response; C-reactive protein; FGF2; MMP8; troponin I; body temperature
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — From each patient 10 ml of venous blood will be collected twice - just before ablation and 24 hours afterwards - and centrifugated to obtain serum.
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate inflammatory response as a prognostic factor of atrial fibrillation recurrency after ablation. Inflammatory response will be assessed by double measurement of C-reactive protein, fibroblast growth factor 2 (FGF2), matrix metallopeptidase 8 (MMP8) and body temperature. Dynamics of change of troponin I will be measured additionally.

After ablation each patient will be monitored with ECG telemonitoring system for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* signed consent;
* criteria for ablation of atrial fibrillation.

Exclusion Criteria:

* previous pulmonary veins isolation;
* ablation other than pulmonary veins isolation during the procedure;
* atrial fibrillation at the beginning of ablation procedure;
* usage of 'single shot' devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study includes adult patients qualified for ablation due to atrial fibrillation.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation within the first 7 days after ablation | within the first 7 days after ablation

SECONDARY OUTCOMES:
Atrial fibrillation within 6 months after ablation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcin D Grabowski, PhD, Study Chair — 1st Department of Cardiology Medical University of Warsaw; Paweł Balsam, PhD, Study Chair — 1st Department of Cardiology Medical University of Warsaw; Piotr Lodziński, PhD, Study Chair — 1st Department of Cardiology Medical University of Warsaw; Grzegorz Opolski, Professor, Study Chair — 1st Department of Cardiology Medical University of Warsaw
Locations (1):
- 1st Department of Cariology of Medcial University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes